CLINICAL TRIAL: NCT07201506
Title: Real-Time Intracardiac Echocardiography for Ventricular Arrhythmia Ablation: A Randomized Controlled Trial
Brief Title: Real-Time Intracardiac Echocardiography for Ventricular Arrhythmia Ablation
Acronym: REAL-ICE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: REAL-ICE
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Ablation of Arrhythmias; Premature Ventricular Contractions; Ventricular Tachycardia; Ventricular Arrhythmia
MeSH Terms: conditions — Ventricular Premature Complexes; Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of SOUNDSTAR® ICE Catheter (Experimental): Use of SOUNDSTAR® ICE Catheter for premature ventricular contraction (PVC) and ventricular tachycardia (VT) ablation
  Interventions: Device: PVC and VT ablation with ICE
- Usual Care: no use of SOUNDSTAR® ICE Catheter (Active Comparator): Usual Care: No use of SOUNDSTAR® ICE Catheter for premature ventricular contraction (PVC) and ventricular tachycardia (VT) ablation
  Interventions: Device: PVC and VT ablation without ICE

INTERVENTIONS:
Device: PVC and VT ablation with ICE — Premature ventricular contraction (PVC) and ventricular tachycardia (VT) ablation with intracardiac echocardiography (ICE)
  Arms: Use of SOUNDSTAR® ICE Catheter
Device: PVC and VT ablation without ICE — Premature ventricular contraction (PVC) and ventricular tachycardia (VT) ablation without intracardiac echocardiography (ICE)
  Arms: Usual Care: no use of SOUNDSTAR® ICE Catheter

SUMMARY:
This study is investigating whether using ultrasound directly inside the heart during ablation of heart rhythm disorders in the ventricles can reduce radiation exposure for patients.

During an ablation, catheters are guided through the heart to treat the abnormal electrical signals. Usually, X-ray imaging (fluoroscopy) is used to see where the catheters are, which exposes both patients and hospital staff to radiation.

The study is randomized and controlled: half of the participants will have the ablation with ultrasound inside the heart, and the other half will have the standard ablation without ultrasound during the procedure. The main goal is to compare the amount of X-ray time used during the procedure. Secondary goals are to look at safety, effectiveness, and the total procedure time.

Patients with premature ventricular contractions or ventricular tachycardia can take part. A total of 70 people will be included, 35 in each group. Using ultrasound inside the heart makes it possible to see the catheters and heart structures directly, so many steps can be done without X-rays. This could make ablations safer and reduce radiation exposure.

The study is being carried out at Inselspital, Bern University Hospital, and at University Hospital Basel. All steps are standardized and data are collected carefully. The results will show whether ultrasound during ablations can significantly reduce radiation and make ablations more efficient and safer.

ELIGIBILITY:
Inclusion Criteria:

* Patients (≥18y) undergoing a premature ventricular contraction or ventricular tachycardia ablation.

Exclusion Criteria:

* Origin of ventricular arrhythmia with high likelihood in the right ventricular outflow tract (left-bundle-inferior axis, >V4 transition precordially)
* Primary epicardial ablation planned
* Congenital heart disease
* Presence of a mechanical tricuspid valve prosthesis
* Unwilling or unable to comply fully with study procedures and followup

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Total fluoroscopy time (minutes) | Day 0 (during procedure)
  Total fluoroscopy time (minutes) from the start to the end of the ablation procedure of ventricular arrhythmias

SECONDARY OUTCOMES:
Dose area product | Day 0 (during procedure)
  Dose area product (cGy·cm²)
Cumulative radiation dose | Day 0 (during procedure)
  Cumulative radiation dose (mGy)
Total procedure time (minutes) | Day 0 (during procedure)
  Procedure start time is defined as the time of first vascular puncture (stick), and procedure end time is defined as the placement of the vascular closure suture.
Rate of acute procedural success | Day 0 (during procedure)
  Defined as a reduction of premature ventricular contraction (PVC) burden by ≥80% and/or ventricular tachycardia (VT) non-inducibility or non-inducibility of clinical VT
Rate of sustained VT during follow-up | Day 0-90 after procedure
  Any sustained ventricular tachycardia episode (lasting ≥30 seconds or requiring an intervention by implantable cardioverter defibrillator). Assessed by a 7-day Holter and/or an implanted cardiac device, if available.
PVC reduction (%) during follow-up | Day 0-90 after procedure
  Reduction of premature ventricular contraction (PVC) burden by ≥80%. Assessed by a 7-day Holter and/or an implanted cardiac device, if available.

OTHER OUTCOMES:
Safety outcome: Rate of serious adverse events related to index ablation | Day 0-90 after procedure
  Composite endpoint of cardiac tamponade requiring drainage, serious vascular complications requiring interventions, stroke/TIA, coronary artery injury requiring intervention, valvular injury requiring intervention, procedural atrioventricular block requiring pacemaker implantation, death after index ablation

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Basel
  - Inselspital, Bern University Hospital, Bern

IPD SHARING:
Plan to Share IPD: Undecided